CLINICAL TRIAL: NCT03908970
Title: A Multicenter, Randomized, Double-blind, Vehicle Controlled, Parallel-group Comparison Trial to Demonstrate the Superiority of 1% OPA-15406 Ointment to the Vehicle in Adult Patients With Atopic Dermatitis (Phase 3 Trial)
Brief Title: Comparison Trial of OPA-15406 Ointment in Adult Patients With Atopic DermatitisSyndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 271-102-00007
Record Dates: First submitted 2019-04-07; First posted 2019-04-09 (Actual); Results first posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — difamilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1% OPA-15406 (Experimental): Twice daily
  Interventions: Drug: 1% OPA-15406
- Placebo (Placebo Comparator): Twice daily
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: 1% OPA-15406 — Twice daily
  Arms: 1% OPA-15406
Drug: Placebos — Twice daily
  Arms: Placebo

SUMMARY:
To demonstrate the superiority of IMP (1% OPA-15406 ointment or vehicle) to the vehicle when administered twice daily for 4 weeks using success rate in Investigator's Global Assessment (IGA) at Week 4 as the primary endpoint in adult patients with AD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AD based on the Japanese Dermatological Association's criteria
* History of AD for at least 3 years
* Atopic dermatitis affecting more than or equal to 5%, to less than or equal to 40% of body surface area (BSA, excluding scalp) at the screening and baseline examinations
* IGA score of 2 or 3 at the screening and baseline examinations

Exclusion Criteria:

* Subjects who have an AD or contact dermatitis flare-up defined as a rapid intensification of AD, within 28 days prior to the baseline examination

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-12-28 (Actual); Study Completion 2019-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Osamu Sato, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Kitago Hifuka Clinic, Sapporo, Japan

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- 1% OPA-15406: Subjects were treated with assigned 1% OPA-15406 ointment twice daily.
- Placebo: Subjects were treated with assigned 0% OPA-15406 ointment twice daily.
Period: Overall Study
Arm/Group | 1% OPA-15406 | Placebo
Started | 182 | 182
Completed | 165 | 135
Not Completed | 17 | 47
Not completed — Adverse Event | 7 | 21
Not completed — Physician Decision | 1 | 4
Not completed — Withdrawal by Subject | 9 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1% OPA-15406 | Placebo | Total
Number analyzed (Participants) | 182 | 182 | 364
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (10.9) | 32.1 (10.6) | 31.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 81 | 167
  Male | 96 | 101 | 197
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 182 | 182 | 364
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 182 | 182 | 364

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate of Investigator's Global Assesment(IGA) of Disease Severity
Description: The investigator or subinvestigator assessed the skin symptoms using IGA. The investigator or subinvestigator scored the severity (0 = clear, 1 = almost clear, 2 =mild, 3 = moderate, 4 = severe/very severe) of the overall symptoms of the treatment area (erythema, infiltration, papules, effusion and scab formation) from baseline to Week 4. Incidence of success in IGA is defined as the rate of subjects whose IGA score is 0 (clear) or 1 (almost clear) and has improved by at least 2 grades (responders) from baseline.
Time Frame: At Week 4
Measure: Number (95% Confidence Interval); unit: percentage of perticipants
Arm/Group | 1% OPA-15406 | Placebo
Number analyzed (Participants) | 182 | 182
percentage of perticipants | 38.46 [31.36 to 45.95] | 12.64 [8.18 to 18.36]

2. Secondary Outcome: Change From Baseline in Eczema Area and Severity Index (EASI) Score
Description: The investigator or sub investigator assessed the symptoms of AD using EASI. EASI's minimum and maximum scores are 0 and 72 scores respectively. The higher the EASI score is, the more severe the symptoms of AD, and a negative change from the baseline means improvement and a positive change means worsening. The investigator or sub investigator scored the severity (0-3 points) and affected BSA (%) based on the 4 symptoms (erythema, infiltration/papules, excoriation, and lichenification) on the 4 body regions (face, neck and head ; upper limbs ;trunk; and lower limbs).
Time Frame: Baseline, Week 4
Population: Number of participants analyzed represents number of participants with data at both Baseline and Week4. Participants who have no data were excluded.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 1% OPA-15406 | Placebo
Number analyzed (Participants) | 166 | 134
score on a scale | -4.17 (0.50) | -0.08 (0.52)

3. Secondary Outcome: Change From Baseline in Verbal Rating Scale (VRS) for Pruritus Score
Description: The investigator or subinvestigator evaluated the pruritus intensity based on VRS. The subjects evaluated the pruritus intensity according to the following criteria. The subjects recorded the level of pruritus and the time and date of evaluation in a pruritus diary.
  0: None
  1. Mild
  2. Moderate
  3. Severe
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 1% OPA-15406 | Placebo
Number analyzed (Participants) | 166 | 134
score on a scale | -0.65 (0.06) | -0.04 (0.07)

ADVERSE EVENTS:
Time Frame: Treatment period (4 weeks)
Arm/Group | 1% OPA-15406 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/182 | 0/182
Serious Adverse Events (participants affected / at risk) | 0/182 | 0/182
Other Adverse Events (participants affected / at risk) | 7/182 | 22/182
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1% OPA-15406 (N=182) | Placebo (N=182)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 7 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT03908970/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT03908970/SAP_001.pdf